CLINICAL TRIAL: NCT03157700
Title: Interactive Technology for Media Literacy Drug Prevention in Community Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Prevention, LLC (Industry)
Collaborators: Rutgers University (Other); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2R42DA039595-02A1 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-17 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Factorial design in which participants are randomly assigned to treatment and control groups. The control is a delayed intervention condition, receiving the intervention after the treatment condition is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL media (Experimental): Participants in this group will be assigned to use the REAL media curriculum.
  Interventions: Behavioral: REAL media curriculum
- Programming as usual (No Intervention): Participants in this group will participate in 4-H programming as usual. They will have the opportunity to use the REAL media curriculum at the conclusion of the study.

INTERVENTIONS:
Behavioral: REAL media curriculum — REAL media is a 5-level, interactive, self-paced, e-learning media literacy curriculum to prevent youth substance use.
  Arms: REAL media

SUMMARY:
This Phase II STTR will evaluate an interactive, self-paced, e-learning media literacy intervention, REAL media, to prevent youth substance use among youth in the 4-H organization. Participating 4-H clubs will be randomly assigned to use the curriculum or continue current practices with the option for delivery at the end of the study. 4-H members (ages 13-15) will complete a pretest, immediate posttest and follow-up posttests at 3 and 9 months to assess effects.

DETAILED DESCRIPTION:
REAL media is an interactive, self-paced, e-learning media literacy curriculum that prevents adolescent substance use among 13-15-year-old teens. The program consists of 5 levels. Levels 1 to 4 are 15-25 minutes; level 5 allots time for message production done offline. Activities lead students to engage in critique and analysis of arguments present/absent from pro-ATOD and other popular product messages and to begin the process of refuting and counter-arguing these messages. These skills are reinforced in level 5 using an active involvement strategy in which youth plan and produce anti-ATOD messages. Users first plan their message via an online worksheet, which requires engagement with and application of media literacy concepts rather than focus exclusively on technology and/or production features. Next, participants design their posters/videos and upload their messages to a social media site as part of a contest, where they recruit peers and family to like or comment on their message.

ELIGIBILITY:
Inclusion Criteria:

* 4-H members and leaders must belong to a participating club in Pennsylvania, Ohio, New Jersey, West Virginia, or Maryland
* members must be between the ages of 13-15
* club leaders must be at least 21 years of age
* written parental consent and assent from members
* written consent from club leaders (online assent)

Exclusion Criteria:

* the inability to speak or read American English
* access to and the ability to use a computer, or navigate the Internet
* for youth, lack of parental consent/youth assent/leader consent

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Change in 15-item Intentions to Use Substances Measure | Change in intentions to use within the next month from baseline to 3 months post baseline.
  Self reported likelihood of using alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana in the following scenarios: at a party, while hanging out with friends, and while by yourself. Response options include Definitely no, No, Yes, and Definitely Yes.
Change in 15-item Intentions to Use Substances Measure | Change in intentions to use within the next month from baseline to 9 months post baseline.
  Self reported likelihood of using alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana in the following scenarios: at a party, while hanging out with friends, and while by yourself. Response options include Definitely no, No, Yes, and Definitely Yes.
Change in 5-item Lifetime Substance Use Measure | Change in lifetime (e.g., ever tried) use from baseline to 3 months post baseline.
  Self reported lifetime use of (e.g., whether you ever tried) alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana. Response options include Yes and No.
Change in 5-item Lifetime Substance Use Measure | Change in lifetime (e.g., ever tried) use from baseline to 9 months post baseline.
  Self reported lifetime use of (e.g., whether you ever tried) alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana. Response options include Yes and No.
Change in 5-item Frequency of Substance Use Measure | Change in frequency of use from baseline to 3 months post baseline.
  Self reported frequency of use of alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana. Response options include range from 0 days to 30+ days.
Change in 5-item Frequency of Substance Use Measure | Change in frequency of use from baseline to 9 months post baseline.
  Self reported frequency of use of alcohol, cigarettes, chewing tobacco (or snuff, dip, snus, or dissolvable tobacco products), e-cigarettes, and marijuana. Response options include range from 0 days to 30+ days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hecht, Ph.D., Principal Investigator — Real Prevention, LLC; Kathryn Greene, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers, The State University of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Once study is completed and publications submitted.

REFERENCES:
- [Derived] Greene K, Choi HJ, Glenn SD, Ray AE, Hecht ML. The Role of Engagement in Effective, Digital Prevention Interventions: the Function of Engagement in the REAL Media Substance Use Prevention Curriculum. Prev Sci. 2021 Feb;22(2):247-258. doi: 10.1007/s11121-020-01181-9. Epub 2020 Nov 3. PMID 33140287
- [Derived] Greene K, Ray AE, Choi HJ, Glenn SD, Lyons RE, Hecht ML. Short term effects of the REAL media e-learning media literacy substance prevention curriculum: An RCT of adolescents disseminated through a community organization. Drug Alcohol Depend. 2020 Sep 1;214:108170. doi: 10.1016/j.drugalcdep.2020.108170. Epub 2020 Jul 10. PMID 32693198